CLINICAL TRIAL: NCT01769157
Title: Single-center, Randomized, Double-Blinded, Comparative Study of the Effectiveness of L-carnitine in Patients'Fatigue Degree Changing With Hypothyroidism Who Take Levothyroxine
Brief Title: Effects of L-carnitine on Hypothyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Principal Investigator, Sin Gon Kim, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LC-TH-1101
Record Dates: First submitted 2013-01-10; First posted 2013-01-16 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-carnitine (Active Comparator): L-carnitine 330mg, 3 tablet twice daily
  Interventions: Drug: L-carnitine
- Placebo (Placebo Comparator): placebo drug, 3 tablet twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-carnitine
  Arms: L-carnitine
Drug: Placebo
  Arms: Placebo

SUMMARY:
L-carnitine and thyroid hormone tended to antagonize reciprocally in human body. Urinary excretion of L-carnitine decreased in hypothyroid patients, and levothyroxine supplementation increased excretion of L-carnitine. The investigators hypothesized that supplying L-carnitine to hypothyroid patients with fatigue symptom could improve the quality of life, and fatigue score in them. Therefore, the investigators planned to compare the efficacy of L-carnitine and placebo in hypothyroid patients who had taken levothyroxine.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypothyroidism with fatigue symptom
* Currently use of the same amount of levothyroxine over at least six months
* Normal serum free T4 level

Exclusion Criteria:

* Current smoker
* Serum hemoglobin level of under 12mg/dL
* Clinical diagnosis of diabetes mellitus or fasting serum glucose level ≥ 126mg/dL or HbA1c level ≥ 6.5%
* History of significant heart failure
* History of large amount of alcohol consumption
* Uncontrolled hypertension (systolic blood pressure ≥ 160 millimeter of mercury (mmHg) or diastolic blood pressure ≥ 100 mmHg
* pregnant, or planning to be pregnant, or breast feeding women
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2 times of normal limit
* serum Cr level > 2.0mg/dL

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity scale | baseline and 12 weeks
  Change from Baseline in Fatigue severity scale at 12 weeks (scoring 'fatigue severity scale' at baseline and 12 weeks)

SECONDARY OUTCOMES:
Wessely and Powell score | baseline and 12 weeks
  Change from Baseline in Wessely and Powell score at 12 weeks (scoring 'Wessely and Powell score' at baseline and 12 weeks)

OTHER OUTCOMES:
thyroid function test | baseline and 12 weeks
  measure thyroid-stimulating hormone and free T4 at baseline and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

REFERENCES:
- [Derived] An JH, Kim YJ, Kim KJ, Kim SH, Kim NH, Kim HY, Kim NH, Choi KM, Baik SH, Choi DS, Kim SG. L-carnitine supplementation for the management of fatigue in patients with hypothyroidism on levothyroxine treatment: a randomized, double-blind, placebo-controlled trial. Endocr J. 2016 Oct 29;63(10):885-895. doi: 10.1507/endocrj.EJ16-0109. Epub 2016 Jul 16. PMID 27432821